CLINICAL TRIAL: NCT00607633
Title: Candesartan and Candesartan/ Hydrochlorothiazide in the Treatment of Patients With Essential Hypertension and a Concomitant Disease Left Ventricular Hypertrophy
Brief Title: Candesartan and Candesartan/ Hydrochlorothiazide in the Treatment of Patients With Hypertension and LVH
Acronym: CandLE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Andrea Pahor, AstraZeneca Germany
Other Study IDs: NIS-CGE-ATA-2007/2
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Last update posted 2008-02-06 (Estimated); Status verified 2008-01

CONDITIONS: Essential Hypertension; Left Ventricular Hypertrophy
Keywords: essential hypertension; ARB; left ventricular hypertrophy; candesartan
MeSH Terms: conditions — Essential Hypertension; Hypertrophy, Left Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patient with essential hypertension and LVH under treatment with candesartan or candesartan HCT

SUMMARY:
The CandLE study with at maximum daily dose of 32 mg candesartan or 16/12.5 mg candesartan/hydrochlorothiazide has the objective to evaluate under naturalistic conditions, i.e. under routine medical care conditions, the impact of the antihypertensive therapy with candesartan or candesartan/HCT on relevant medical parameters related to the left ventricular hypertrophy (LVH) as well as the efficacy and tolerability of candesartan or candesartan/HCT in subjects suffering from essential hypertension..

ELIGIBILITY:
Inclusion Criteria:

* essential hypertension
* left ventricular hypertrophy
* under candesartan treatment

Exclusion Criteria:

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Ambulant patient
Sampling Method: Probability Sample
Enrollment: 686 (Actual)
Dates: Start 2007-01; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
to estimate under naturalistic conditions the impact of the antihypertensive therapy with candesartan or candesartan/HCT on pre-post change from Visit 1 to Visit 2 of Sokolow-Lyon index, Cornell index and Left Ventricular Mass Index. | app. 3 monthly

SECONDARY OUTCOMES:
to estimate the change of the systolic and diastolic blood pressure, separately by the (maximum) prescribed daily dose of candesartan or candesartan/ HCT | app. 3 monthly
to gain further insight into the occurrence of unknown, unexpected and/or rarely occurring adverse events (AE) by estimating the incidence under naturalistic conditions. | app. 3 monthly

CONTACTS AND LOCATIONS:
Overall Officials: F. Sonntag, MD, Principal Investigator — Cardiologist, Henstedt-Ulzburg; Andrea Pahor, MD, Study Chair — MED Dep., AstraZeneca Germany